CLINICAL TRIAL: NCT07199777
Title: A Phase 2a, Randomized, Double-masked, Placebo-controlled, Multicenter Study to Evaluate the Safety, Tolerability, and Efficacy of SNP318 in Patients With Diabetic Macular Edema
Brief Title: A Phase 2a Study to Evaluate the Safety, Tolerability, and Efficacy of SNP318 in DME Patients
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: SciNeuro (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SNP318-102
Record Dates: First submitted 2025-09-22; First posted 2025-09-30 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Diabetic Macular Edema; DME

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- SNP318 (Experimental)
  Interventions: Drug: SNP318
- Matching Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SNP318 — Once daily, oral administration
  Arms: SNP318
Drug: Placebo — Once daily, oral administration
  Arms: Matching Placebo

SUMMARY:
The objective of this study is to assess the safety, efficacy, and tolerability of SNP318 in patients with DME.

DETAILED DESCRIPTION:
DME is a prevalent complication of diabetic retinopathy, resulting in fluid accumulation in the macula due to the leakage of fluid from damaged retinal blood vessels. It is a leading cause of vision impairment in diabetic patients and can significantly affect quality of life if left untreated. SNP318 is a small molecule and selective inhibitor of Lp-PLA2. It plays a critical role in the regulation of the pro-neuroinflammatory pathway, which is implicated in the pathogenesis of multiple diseases.

This is a phase 2a, randomized, double-masked, placebo-controlled, multicenter study to evaluate the safety, tolerability, and efficacy of SNP318 in patients with Diabetic Macular Edema. Participants who consent will undergo a 3-week screening period to evaluate their eligibility. Once enrolled, participants will be randomized to receive orally either SNP318 or placebo for up to 12 weeks, and then enter into a 4-week follow up period.

ELIGIBILITY:
Main Inclusion Criteria:

1. Confirmed diabetes mellitus Type 1 or Type 2, with stable glycemic control
2. Center-involved DME with CST >=320 µm (Study eye)
3. BCVA between 82 and 25 letters, inclusive (Study eye)
4. BCVA score ≥ 25 letters (Non-study eye)

Main Exclusion Criteria:

1. Use of the last intravitreal anti-VEGF injection in the study eye within 90 days prior to Screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Safety Events | 12 weeks
  Incidence of adverse events (AEs) / serious adverse events (SAEs)
Central Subfield Thickness (CST) | 12 weeks
  Spectral Domain Optical Coherence Tomography (SD-OCT) measurements of CST

SECONDARY OUTCOMES:
Visual Acuity | 12 weeks
  Best Corrected Visual Acuity (BCVA) assessed according to ETDRS criteria
Pharmacokinetics (PK) | 12 weeks
  Plasma concentrations of SNP318
Pharmacodynamics | 12 weeks
  Plasma Lp-PLA2 activity